CLINICAL TRIAL: NCT04169256
Title: A Phase I, Single Centre, Randomized, Double-blinded, Placebo-controlled, Single Ascending Dose-Escalation, Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profile of HYR-PB21 and Liposome Bupivacaine in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profile of HYR-PB21 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fruithy Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HYR-PB21-AU-01
Record Dates: First submitted 2019-11-06; First posted 2019-11-19 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Acute Postoperative Pain
Keywords: pain; postoperative; local anesthesia; long-action
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HYR-PB21 & Placebo (Experimental)
  Interventions: Drug: HYR-PB21; Other: Normal Saline
- Liposome Bupivacaine & Placebo (Active Comparator)
  Interventions: Drug: Liposomal bupivacaine; Other: Normal Saline

INTERVENTIONS:
Drug: HYR-PB21 — HYR-PB21 for injection 100mg, 200mg,or 400mg by single subcutaneous injection on the abdomen
  Arms: HYR-PB21 & Placebo
Drug: Liposomal bupivacaine — Liposome Bupivacaine Suspension for injection 200mg by single subcutaneous injection on the abdomen
  Arms: Liposome Bupivacaine & Placebo
Other: Normal Saline — Normal Saline 30ml, or 40mL by single subcutaneous injection on the abdomen

SUMMARY:
This study is the first time into human study (FTIH) for HYR-PB21 for injection. The study will evaluate the safety, pharmacokinetics (PK) and pharmacodynamics (PD) of single ascending and single subcutaneous dose of HYR-PB21 for injection in healthy adult volunteers.The results of this study are intended to be used to identify appropriate and well tolerated doses of HYR-PB21 for injection to be used in further studies. A comparison of PK/PD characteristics between HYR-PB21 for injection and EXPAREL will also be included in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provide written informed consent.
2. Subjects who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
3. Subjects with liver function tests (LFTs) within the reference range, or deemed clinically not significant by the investigator or delegate.
4. Male or female (of non-child bearing potential) between 18 and 50 years of age, inclusive.
5. If female, be of non-childbearing potential: e.g. post-menopausal for ≥12 consecutive months with follicle stimulating hormone (FSH) ≥40 mIU/mL at Screening; or surgical sterilization for at least 90 days prior to screening e.g., tubal ligation or hysterectomy. Note: Provision of documentation is not required for female sterilization, verbal confirmation is adequate.
6. Male patients must be surgically sterile (biologically or surgically) or commit to the use of a reliable method of birth control for the duration of the study until at least 30 days after the administration of study medication.
7. Have a body mass index 18-30 kg/m2 (inclusive).
8. Blood pressure < 140/90 mmHg at screening and heart rate <100 bpm. One repeat assessment is permitted. Screening laboratory tests that are deemed to be non-clinically significant by the investigator.
9. Subjects must not have donated or lost more than 400 mL of blood within 12 weeks of dosing, more than 200mL of blood within 4 weeks of dosing or donated any blood within 2 weeks of dosing.
10. Subjects must not donate sperm or egg during study or in 30 days after dosing.
11. Be able to understand the study procedures, comply with all study procedures, and agree to participate in the study program.
12. Be able to understand and communicate in English.

Exclusion Criteria:

1. History of hypersensitivity or idiosyncratic reactions to amide-type local anaesthetics.
2. History of abnormal bleeding tendencies/clotting disorders.
3. History of glucose-6-phosphate dehydrogenase (G6PD) deficiency.
4. History of significant neurological, hepatic, renal, endocrine, cardiovascular, cardiac arrhythmias, gastrointestinal, pulmonary, or metabolic disease.
5. Regular use of anticoagulants.
6. Received any investigational drug within 30 days or 5 half-lives of the investigational drug prior to study drug administration, and/or has planned administration of another investigational product or procedure during his/her participation in this study.
7. Currently pregnant or nursing.
8. The subject has a history of substance abuse or smoking, a positive ethanol breath test, urine cotinine, or urine drug screen at screening or at check-in. One repeat test is allowable if a false positive is suspected at the investigator's discretion.
9. The subject has a positive serum hepatitis B surface antigen or positive HCV antibody test at the Screening Visit.
10. Subject has a positive HIV test at the Screening Visit.
11. Received bupivacaine, other local anaesthetic, prescription or OTC medications, herbal remedies or supplements per standard practice within 14 days of first study drug administration. Received caffeine and alcohol consumption within 48 h prior to drug administration.
12. Any conditions, that according to investigator's best judgment, prevent participation in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration-versus-time curve from the time of administration to the time of the last quantifiable concentration calculated using the log-linear trapezoidal rule | 15 days
  Pharmacokinetic parameters will be estimated from plasma bupivacaine measurements using non-compartmental analysis, based on the sampling schedule at predose (on Day 1 prior to study drug administration); 0.25, 0.5, 1, 2, 4, 8, 12, 18, 24, 30, 36, 48, 60, 72, 96, 120, 144, 168 hours and 14 days post-dose.
The area under the plasma concentration-versus-time curve from the time of administration extrapolated to infinity. | 15 days
  The residual area from the time of the last quantifiable concentration to infinity is to be calculated using the approximation
The maximum observed plasma bupivacaine concentration obtained directly from the experimental data without interpolation. | 15 days
The time to maximum plasma concentration (Cmax) | 15 days
The apparent terminal elimination half-life calculated as 0.693/λz | 15 days
The apparent terminal elimination rate constant determined by log-linear regression of the terminal log-linear segment of the plasma concentration-versus-time curve | 15 days
The average Von Frey filament pressure across five test points at each protocol scheduled time-point | 8 days
  Detection of the loss of feeling at injection site (at selected five representative test points) by Von Frey filaments in different pressures will be estimated at 15-45 min pre-dose; 0.25, 0.5 , 1, 2, 4, 8, 12, 18, 24, 30, 36, 48, 60, 72, 96, 120, 144, and 168 hour post-dose.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | 15 days
Investigator assessment of the ECG (normal, abnormal - not clinically significant, abnormal - clinically significant) | 15 days
  12-lead ECG will be obtained at screening, check-in，15-45 min pre-dose;0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 168 hours,and 14 days post-dose using an ECG machine for measurements of PR, QRS, QT, QTcF intervals,and heart rate.
Observer's assessment of alertness/sedation(OAA/S) scale | 5 days
  Six categories of responsiveness scores were characterized by the following responses for the OAA/S assessment:
  * Responds readily to name spoken in normal tone (5 scores)
  * Responds lethargically to name spoken in normal tone (4 scores)
  * Responds only after name is called loudly, repeatedly, or both (3 scores)
  * Responds only after mild prodding or shaking (2 scores)
  * Responds only after painful trapezius squeeze (1 score)
  * Does not respond to painful trapezius squeeze (0 score)

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, Southwest, Australia

IPD SHARING:
Plan to Share IPD: No